CLINICAL TRIAL: NCT07265154
Title: Gait Training in Above Knee Amputation Patients Using Artificial Intelligence
Brief Title: Gait Training and Artificial Intelligence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Collaborators: Badr University (Other); Benha University (Other); Al Salam University (Other)
Responsible Party: Principal Investigator, Mohammed E. Ali, Lecturer of Physical Therapy, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/004661
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Above Knee Amputation; Amputation
Keywords: Amputation; Above Knee Amputation; Artificial Intelligence; Gait training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Gait Training Using Artificial Intelligence
  Interventions: Device: Artificial Intelligence
- group B (No Intervention): Traditional Physical Therapy Program

INTERVENTIONS:
Device: Artificial Intelligence — using artificial intelligence in gait training for above knee amputee
  Arms: group A

SUMMARY:
Effect of Using Artificial Intelligence on Gait Training in Above Knee Amputation Patients

ELIGIBILITY:
Inclusion Criteria:

* All patients have above-knee amputations.
* All patients have no other neurological diseases affecting gait.
* All patients have no other neurological diseases affecting muscle balance.
* All patients have no other complications affecting joint ROM.

Exclusion Criteria:

* Patients have any complications affecting joint ROM.
* Patients have any neurological condition affecting muscle balance.
* Patients have any neurological condition affecting gait.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Medio-lateral Stability Index (MLSI) | Day 0, Day 30
  Medio-lateral Stability Index (MLSI) represents fluctuations from the horizontal around the mediolateral axis
Anterior-posterior Stability Index (APSI) | Day 0, Day 30
  Anterior-posterior Stability Index (APSI) represents fluctuations from the horizontal around the anteroposterior axis
Overall Stability Index (OSI) | Day 0, Day 30
  Overall Stability Index (OSI) a composite of MLSI and APSI so it is sensitive to changes in both directions

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy,, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hartley H, Cassidy E, Bunn L, Kumar R, Pizer B, Lane S, Carter B. Exercise and Physical Therapy Interventions for Children with Ataxia: A Systematic Review. Cerebellum. 2019 Oct;18(5):951-968. doi: 10.1007/s12311-019-01063-z. PMID 31392562
- [Result] Tatla SK, Radomski A, Cheung J, Maron M, Jarus T. Wii-habilitation as balance therapy for children with acquired brain injury. Dev Neurorehabil. 2014 Feb;17(1):1-15. doi: 10.3109/17518423.2012.740508. Epub 2012 Dec 11. PMID 23231377
- [Result] 1. Nehad A. Abo-Zaid, Nesma A Helmy, Nader I Elsayed, Amira H Mohammed. Wii Sport versus task-oriented training on gait in unilateral cerebral palsy: A randomized controlled trial. Conference: Journal of Human Sport and Exercise. Autumn Conferences of Sports Science2021.16. Proc2.36, doi: 10.14198/jhse.
- [Result] Abo-Zaid NA, El-Gendy AM, Hewidy I, Essam Ali M, Sabbahi A. Influence of aerobic exercise on inhibitory control of executive functions in children with hemiplegic cerebral palsy: A randomized controlled trial. Clin Rehabil. 2024 Mar;38(3):337-346. doi: 10.1177/02692155231208578. Epub 2023 Oct 26. PMID 37885221
- [Result] 27. Nehad A Abo-zaid, Hebatallah M Zaghloul, Heba A Khalifa., Mohammed E Ali, Mohamed Y Abdelsamee. Efficacy of Lower Extremity Mirror Therapy on Balance in Children with Hemiplegic Cerebral Palsy: A Randomized Controlled Trial International Journal of Psychosocial Rehabilitation, 2020, Vol. 24, Issue 08
- [Result] Nolan L, Grigorenko A, Thorstensson A. Balance control: sex and age differences in 9- to 16-year-olds. Dev Med Child Neurol. 2005 Jul;47(7):449-54. doi: 10.1017/s0012162205000873. PMID 15991864
- [Result] Kitago T, Krakauer JW. Motor learning principles for neurorehabilitation. Handb Clin Neurol. 2013;110:93-103. doi: 10.1016/B978-0-444-52901-5.00008-3. PMID 23312633
- [Result] Dewar R, Love S, Johnston LM. Exercise interventions improve postural control in children with cerebral palsy: a systematic review. Dev Med Child Neurol. 2015 Jun;57(6):504-20. doi: 10.1111/dmcn.12660. Epub 2014 Dec 18. PMID 25523410
- [Result] 45. Rafaela Ribeiro da Silva, Cristina Iwabe-Marchese. Using virtual reality for motor rehabilitation in a child with ataxic cerebral palsy: case report. Fisioter Pesq. 2015; 22(1):97-102, doi.org/10.590/1809-2950/13375322012015